CLINICAL TRIAL: NCT04868227
Title: Scottish Vitamin D Intervention Study
Acronym: (SCoViDS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: Cancer Research UK (Other); Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2014/0058
Record Dates: First submitted 2021-04-25; First posted 2021-04-30 (Actual); Results first posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: GENE EXPRESSION; Colorectal Cancer
Keywords: VITAMIN D
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: SINGLE GROUP INTERVENTION STUDY
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- INTERVENTION STUDY (Experimental): TREATED WITH 3200IU FULTIUM VITAMIN D3
  Interventions: Dietary Supplement: FULTIUM D3 VITAMIN D3

INTERVENTIONS:
Dietary Supplement: FULTIUM D3 VITAMIN D3 — VITAMIN D3 SUPPLEMENT

SUMMARY:
AIMS To identify the underlying mechanism by which Vitamin D reduces colorectal cancer risk.

OBJECTIVES To demonstrate the effects of vitamin D supplementation on serum vitamin D levels.

To demonstrate dynamic changes in gene expression in response to vitamin D. To demonstrate the mechanism underlying the gene-environment interaction of vitamin D, susceptibility genetic variants (risk genes) and colorectal cancer.

DETAILED DESCRIPTION:
Through National Health Service (NHS) clinical services in colorectal surgery and oncology, patients will be identified and recruited from surgical wards or surgical/oncology out-patient clinics. A sample of participants with and without a new or previous diagnosis of colorectal cancer will be included for comparison.

Participation will consist of two events in the majority of participants. Firstly a in the surgical ward or clinic lasting no longer than 20 minutes in which the research will be discussed and informed consent gained. A blood sample will be taken prior to the conclusion of recruitment and a rectal biopsy taken using a rigid sigmoidoscopy which may or may not be required as part of their routine clinical assessment. Participants will be asked to take pharmaceutical grade vitamin D tablets for 3 months. After 12 weeks of vitamin D supplementation, a final blood sample and rectal biopsy will be taken.

If patients would like to contribute but cannot or would prefer not to take vitamin D, or cannot return for future sampling, a single sampling will be offered. This participant would undergo blood sampling and rectal biopsy as above. After this no further events would occur.

ELIGIBILITY:
Inclusion Criteria:

* Aged 16 years or over.
* Resident of the United Kingdom

Exclusion Criteria:

1. The inability to provide informed consent.
2. Under the age of 16 years.
3. A non-UK resident.
4. Patients who may be at increased risk from rigid sigmoidoscopy:

   * Individuals who are taking anti-coagulation medication.
   * Individuals with platelet disease or other bleeding issues.
   * Individuals with a history of a significant rectal bleed.
   * Suspected or known bowel perforation
   * Anal stenosis
   * Acute peritonitis
   * Colonic necrosis
   * Toxic megacolon
   * Acute severe diverticulitis
   * Diverticular abscess
   * Recent colonic surgery
   * Anal fissure
   * Severe coagulopathy
   * Anticoagulant therapy
   * Severe thrombocytopenia
   * Severe neutropenia
5. Patients who may be at increased risk from Vitamin D supplementation would not be included in the intervention arm but could still be included in the single sample arm:

   * Kidney disease
   * High levels of calcium in the blood
   * Atherosclerosis
   * Sarcoidosis
   * Histoplasmosis
   * Over-active parathyroid gland (hyperparathyroidism)
   * Lymphoma
   * Currently taking thiazide diuretics, digoxin or other cardiac glycosides
   * Known allergy to nuts ( as peanut oil contained within vitamin D preparations)
   * Female subjects of child bearing age who are not taking effective contraception during the period of the trial
6. Patients in whom vitamin D levels may be unpredictable

   * Individuals already established on supplementary Vitamin D.
   * Individuals recently returned to the UK from an overseas holiday.
   * Individuals who have recently lived abroad.
   * Patients on anti-epileptic medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-03-28 (Actual); Primary Completion 2016-04-11 (Actual); Study Completion 2016-07-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm G Dunlop, MD, Principal Investigator — MRC HGU University of Ediniburgh
Locations (1):
- Western General Hospital, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Transcript profiling: Available at https://www.ncbi.nlm.nih.gov/geo/ Gene Expression Omnibus (GEO) identifier (ID) GSE157982. Full phenotypic data available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: AS REQUESTED
Access Criteria: Full protocol and Full phenotypic data available from the corresponding author on reasonable request.

REFERENCES:
- See also: GEO ID GSE157982. — http://www.ncbi.nlm.nih.gov/geo/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Analyses were intended to be conducted irrespective of previous diagnosis status. i.e. Results are not compared between those with/ without previous history of colorectal cancer.
Groups:
- INTERVENTION STUDY (Single Arm Study): TREATED WITH 3200IU FULTIUM VITAMIN D3
  FULTIUM D3 VITAMIN D3: VITAMIN D3 SUPPLEMENT
  Analyses were intended to be conducted irrespective of previous diagnosis status. i.e. Results are not compared between those with/ without previous history of colorectal cancer.
Period: Overall Study
Arm/Group | INTERVENTION STUDY (Single Arm Study)
Started | 50
Completed | 48
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Recruited patients were those both with and without previous history of cancer. However, analyses were intended to be conducted irrespective of previous diagnosis status. i.e. Results are not compared between those with/ without previous history of colorectal cancer.
Arm/Group | INTERVENTION STUDY
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 66 [24 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 26
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Genes Significantly Associated With 25OHD Blood Vitamin D Level
Description: RECTAL MUCOSA GENE EXPRESSION (HT12 microarray. No units on gene expression array)
Time Frame: AT BASELINE
Population: as for baseline characteristics
Measure: Number; unit: significant probes (P<0.01)
Units Other Than Participants: Gene expression HT12 microarray.
Arm/Group | INTERVENTION STUDY
Number analyzed (Participants) | 48
Number analyzed (Gene expression HT12 microarray.) | 47231
significant probes (P<0.01) | 629

2. Primary Outcome: GENE EXPRESSION CHANGE
Description: RECTAL MUCOSA GENE EXPRESSION. We tested supplemented patients (i.e. response to supplementation) for enrichment of the candidate gene-set. Directional gene-set testing was performed in R, using the gene-setTest function in the 'limma' package. We performed participant-level gene-set enrichment testing with a 'response' to supplementation defined as enrichment (P<0.001) of the candidate gene-set after supplementation.
Time Frame: AFTER 12 WEEK'S SUPPLEMENTATION
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | INTERVENTION STUDY
Number analyzed (Participants) | 48
Participants | 9

3. Secondary Outcome: VITAMIN D STATUS
Description: Blood vitamin D level (25-hydroxy-vitamin D (25-OHD) level (nmol/l)) using Liquid chromatography tandem mass spectrometry (LC- MS/MS)
Time Frame: AT BASELINE
Population: Fifty subjects were administered 3200IU/day oral vitamin D3 and matched blood/mucosa resampled after 12 weeks'. Analyses were intended to be conducted irrespective of previous diagnosis status. i.e. Results are not compared between those with/ without previous history of colorectal cancer.
Measure: Median (Inter-Quartile Range); unit: nmol/l
Units Other Than Participants: Plasma
Arm/Group | INTERVENTION STUDY
Number analyzed (Participants) | 50
Number analyzed (Plasma) | 98
nmol/l | 40 [22.5 to 58.5]

4. Secondary Outcome: VITAMIN D STATUS CHANGE
Description: Blood vitamin D level (25-hydroxy-vitamin D (25-OHD) level (nmol/l))
Time Frame: AFTER 12 WEEK'S SUPPLEMENTATION
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: nmol/l
Arm/Group | INTERVENTION STUDY
Number analyzed (Participants) | 50
nmol/l
  Vitamin D Level at Baseline | 35.85 [23.14 to 54.41]
  Vitamin D Level at 12 weeks | 89 [72.25 to 105.75]

ADVERSE EVENTS:
Groups:
- INTERVENTION STUDY: TREATED WITH 3200IU FULTIUM VITAMIN D3. THERE ARE NO INDIVIDUAL ARMS TO REPORT.
  FULTIUM D3 VITAMIN D3: VITAMIN D3 SUPPLEMENT
  Participants were followed up for adverse events for the duration of the study (i.e. during vitamin D treatment) but not beyond.
Arm/Group | INTERVENTION STUDY
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

LIMITATIONS AND CAVEATS:
This intervention study is larger than many published studies of gene expression and vitamin D supplementation, yet may still have limited power to achieve individual gene significance. Unmeasured variation in environmental exposures (e.g. diet or UVB exposure) may have influenced responses,

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes